CLINICAL TRIAL: NCT04641910
Title: Validation Study of a New Cytokine-based Dynamic Stratification Based on FLt3 Ligand Plasma Concentration Kinetic Profile and IL-6 Concentration During Induction of Acute Myeloid Leukemia
Acronym: FLAMVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0406
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples at day 1, day 8, day 15, day 22, day 30
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators have recently demonstrated the strong impact in terms of survivals of Fms-like tyrosine kinase 3 ligand (FL) levels evaluated during intensive induction in acute myeloid leukemia (AML) patients. Indeed, three FL kinetic profiles were delineated: i) sustained increase of FL concentrations between day (D) 1 and D22 (FLI group, n=26, good-risk), ii) increase from D1 to D15, then decrease at D22 (FLD group, n=22, intermediate-risk) and iii) stagnation of low levels (<1000 pg/mL, FLL group, n=14, high-risk). However, with longer follow-up, the investigators have observed that FLI and FLD shared similar outcomes while FLL sub-group kept a very bad prognostic.

Because serum samples from this previous study (called the FLAM/FLAL study) had been frozen-stored, the investigators were able to conduct an ancillary study assessing the potential impact of the kinetics of 6 other cytokines: TNFalpha, stem-cell factor, IL-1beta, IL-6, IL-10 and granulocyte-monocyte colony-stimulating factor (GM-CSF).. Only Il-6 level at D22 (< or >15.5 pg/mL) was associated with outcome allowing to distinguish between higher and lower survivals within the combined FLI/FLD sub-group.

A new prognostic risk-stratification can thus be proposed as follows: FLI/FLD with IL-6 <15.5 pg/mL (favorable), FLI/FLD with IL-6 >15.5 pg/mL (intermediate) and FLL (high-risk).

The aim of this new FLAMVAL study is to validate prospectively in a larger and independent cohort this prognostic risk-stratification i.e. that kinetic profile of FLT3L plasma level from D1 to D22 and Il6 plasma level at day 22 during induction of AML patients are predictive of overall and disease free survivals.

For that purpose, 201 newly diagnosed AML patients treated intensively in the 25 centres of the French Innovative Leukemia Organisation (FILO) will be included in the FLAMVAL study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Confirmed diagnosis of AML according to World Health Organization (WHO) 2016 classification (Arber et al., 2016)
* Non previously treated AML (first-line therapy)
* Patients eligible to standard 3+7 induction chemotherapy with a minimum of 3 days of daunorubicin at 45mg/m2/day or a minimum of 5 days of idarubicin at 8mg/m2/day and a minimum of 7 days of cytarabin at 100mg/m2/day
* Patients receiving any "third drug" combined to the "3+7" scheme, i.e. lomustine, corticotherapy, elthrombopag, gemtuzumab-ozogamycin, any FLT3 inhibitors… are eligible
* Patients receiving CPX-351 (Vyxeos ®) are eligible
* Patients requiring leukapheresis are eligible
* Signed informed consent

Exclusion Criteria:

* Patients diagnosed with Acute Promyelocytic Leukemia (AML-3)
* Adults under guardianship, subjects under protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any newly diagnosed AML patients treated intensively in centres belonging to the FILO group will be eligible for the FLAMVAL study.
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-06-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Confirm that the combination of the kinetic profile of FLT3L plasma levels and the IL-6 plasma level at day22 during induction in AML patients is predictive of overall survival. | 2 years
  time from day 1 of induction to the date of death or of last follow-up
Confirm that the combination of the kinetic profile of FLT3L plasma levels and the IL-6 plasma level at day22 during induction in AML patients is predictive of overall survival. | 2 years
  serum FL concentration is measured at day 1, 8, 15 et 22 of induction by ELISA
Confirm that the combination of the kinetic profile of FLT3L plasma levels and the IL-6 plasma level at day22 during induction in AML patients is predictive of overall survival. | 2 years
  level of IL-6 at day 22 has been also shown to have prognostic impact for FLD/FLI patients

SECONDARY OUTCOMES:
Confirm that the new FL/IL6 risk-model predicts leukemia free survival in first-line AML patients. | 2 years
  Progression-free survival (PFS): time from day 1 of induction to refractory disease or relapse censored at the date of death or last follow-up
Compare the prognostic impact of the new FL/IL6 risk-model with the impact of other parameters known to predict outcome in AML | 2 years
  Refractory status after induction
Study the impact of the new FL/IL6 risk-model in FLT3 ITD or TKD patients receiving or not FLT3 inhibitors | 2 years
  cytokines plasma levels
Study Immune reconstitution during induction | 2 years
  By flow cytometry

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Strasbourg University Hospital, Strasbourg, Bas-Rhin
  - Paoli-Calmette Institute, Marseille, Bouches-du-Rhône
  - Besançon University Hospital, Besançon, Doubs
  - Brest University Hospital, Brest, Finistère
  - Nîmes University Hospital, Nîmes, Gard
  - Bordeaux University Hospital, Bordeaux, Gironde
  - Mulhouse Hospital Center, Mulhouse, Haut-Rhin
  - Toulouse University Cancer Institute, Toulouse, Haute-Garonne
  - Béziers Hospital Center, Béziers, Hérault
  - Montpellier University Hospital, Montpellier, Hérault
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Grenoble University Hospital, Grenoble, Isère
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Angers University Hospital, Angers, Maine-et-Loire
  - Reims University Hospital, Reims, Marne
  - Nancy University Hospital, Nancy, Meurthe-et-Moselle
  - Mercy Regional Hospital, Metz, Moselle
  - Saint-Etienne University Hospital, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Clermont-Ferrand University Hospital, Clermont-Ferrand, Puy-de-Dôme
  - Basque coast hospital center, Bayonne, Pyrénées-Atlantiques
  - Saint-Jean Hospital Center, Perpignan, Pyrénées-Orientales
  - Lyon University Hospital, Lyon, Rhône
  - AP-HP Cochin Hospital, Paris
  - Poitiers University Hospital, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided